CLINICAL TRIAL: NCT07290062
Title: A Phase 1, Multicenter, Open-label, Dose-Finding Study to Investigate the Safety and Pharmacodynamics of a Single Intrathecal Injection of INS1202 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: A Study to Investigate the Safety and Pharmacodynamics of a Single Intrathecal Injection (IT) of INS1202 in Participants With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ARMOR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Gene Therapy LLC (Industry)
Responsible Party: Sponsor
Organization: Insmed Incorporated (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INS1202-101
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Participants with sporadic amyotrophic lateral sclerosis (sALS) will be administered INS1202, IT injection at dose level 1 on Day 1.
  Interventions: Genetic: INS1202
- Cohort 2 (Experimental): Participants with either sALS or SOD1-ALS, will be administered INS1202 via IT injection at dose level 2 on Day 1.
  Interventions: Genetic: INS1202
- Cohort 3 (Experimental): Participants with either sALS or SOD1-ALS, will be administered INS1202 via IT injection at dose level 3 on Day 1.
  Interventions: Genetic: INS1202

INTERVENTIONS:
Genetic: INS1202 — Suspension for injection.

SUMMARY:
The primary objective of this dose-finding study is to evaluate the safety, tolerability and pharmacodynamics of single dose of INS1202 via IT administration in participants ≥ 18 to <80 years of age with ALS who carry superoxide dismutase type 1 (SOD1) mutations or harbor no known ALS-related genetic mutation.

ELIGIBILITY:
Key Inclusion Criteria: -

* Participant with body mass index (BMI) ≥18 kilograms per square meter (kg/m^2).
* Participant with symptomatic ALS as diagnosed by Gold Coast diagnostic criteria.
* Sporadic ALS cohorts: Negative testing for known monogenic mutations associated with familial ALS.
* SOD1-ALS (Cohorts 2 and 3 only): Confirmed pathogenic SOD1 mutation, with negative testing for other genetic mutations associated with familial ALS.
* Any polymorphism or mutation in the coding region will require additional review by the Sponsor to determine compatibility with the study intervention.
* Baseline ALSFRS-R ≥ 24.
* ALS disease duration ≤ 42 months.

Key Exclusion Criteria: -

* Previous treatment for ALS with cellular or gene therapies.
* Any investigational medication or treatment (for ALS or other condition).

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Up to 48 weeks

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of INS1202-101 | Up to 48 weeks
Viral Vector Shedding Following the IT Administration of INS1202 by Droplet Digital Polymerase Chain Reaction (ddPCR) | Baseline, Week 1, Week 2, Week 4, Week 16 and Week 32

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No